CLINICAL TRIAL: NCT05368129
Title: Safety and Efficacy of POT PTCA Balloon Dilatation Catheter for the Optimal Dilation After Drug-eluting Stent Implantation: a Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: Safety and Efficacy of POT PTCA Balloon Dilatation Catheter for the Optimal Dilation After DES Implantation
Acronym: POT-DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President of Nanjing First Hospital, Director of Cardiovascular Department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFH20220425
Record Dates: First submitted 2022-04-25; First posted 2022-05-10 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POT group (Experimental): A total of 24 patients are assigned to POT group after randomization schedule.
  Interventions: Procedure: Balloon dilation
- NCB group (Active Comparator): A total of 24 patients are assigned to NCB group after randomization schedule.
  Interventions: Procedure: Balloon dilation

INTERVENTIONS:
Procedure: Balloon dilation — Balloon dilation was performed after DES implantation.

SUMMARY:
The objective of this randomized control trial is to gain clinical insight on the use of POT PTCA balloon dilatation catheter for the optimal dilation after drug-eluting stent implantation.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the change in minimal stent area (MLA) of POT PTCA balloon dilatation catheter on patients with drug-eluting stent (DES) implantation. Based on the previous studies, the MLA in the proximal and distal 3mm segments was 7.38 mm^2 and 8.08 mm^2 before non-compliant balloon (NCB) dilation, respectively. After NCB dilation, that MSA in the proximal and distal 3mm segments was 7.53mm^2 and 9.55mm^2, respectively. As a result, a total of 48 patients with DES implantation are randomized at a ratio of 1:1 to either POT PTCA balloon dilatation catheter group (POT group) or Quantum Maverick balloon catheter group (NCB group) using a randomization schedule blocked by site.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Men and women 18 years and older;
3. Patients with asymptomatic myocardial ischemia, stable or unstable angina, or acute myocardial infarction with symptoms lasting more than 12 hours;
4. The target lesions was de novo lesion;
5. Reference vessel diameter of target lesion is between 2.25-4.0mm, and the lesion length is less than 15mm(visual inspection);
6. Diameter stenosis of target lesion diameter ≥70% or ≥50%(visual) with ischemia evidence;
7. DES was successfully implanted in target lesions;
8. TIMI 3 blood flow of target vessel before post-dilation.

Exclusion Criteria:

1. Subjects had clinical symptoms and/or ECG changes consistent with ST-elevation myocardial infarction within 12 hours;
2. Allergies to concomitant medications required by the balloon/stent system or protocol used in the study;
3. Cannot tolerate dual antiplatelet therapy;
4. Life expectancy is less than 6 months;
5. Pregnant or lactating women;
6. Participating in another clinical trial and has not completed the primary endpoint observation of the trial;
7. Planned multiple operations, failed to follow the treatment prescribed in the protocol or affected data analysis and interpretation;
8. Restenosis disease;
9. Target lesions with severe calcification require rotary grinding treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Minimal stent area | through PCI procedure completion
  The change of minimum stent area measured by intravascular ultrasound.

SECONDARY OUTCOMES:
PCI success | up to 7 days
  Successful PCI was defined as diameter stenosis of the target lesion ≤30%, no intraprocedure death, Q-wave or non-Q-wave myocardial infarction, or emergency coronary artery bypass grafting.
Device success | through PCI procedure completion
  Success of the device (successful balloon expansion) must meet the following conditions:
  1. Successfully complete the process of delivery, expansion, retraction and withdrawal;
  2. There was no balloon related vascular perforation, C-type or above dissection with limited blood flow, and TIMI grading was not lower than before balloon dilation.

OTHER OUTCOMES:
Death | up to 7 days
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 days
Dissection | through PCI procedure completion
  Vessel dissection was noted during the procedure.
Stent thrombosis | Within 24 hours after PCI
  Stent thrombosis occurred within 24 hours after PCI.
Perioperative myocardial infarction | Within 48 hours after PCI
  Perioperative myocardial infarction within 48 hours after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No